CLINICAL TRIAL: NCT00071578
Title: Comparison of Dialectical Behavior Therapy and Supportive Therapy for Binge Eating Disorder
Brief Title: Comparing Two Group Therapy Treatments for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Debra L. Safer, Asst professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23MH066330 (NIH); K23MH066330 (NIH); DSIR 8K-RTAT
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Eating Disorders
Keywords: Psychotherapy; Treatment
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group therapy Negative Emotion Focus
  Interventions: Behavioral: Group Psychotherapy-Negative Emotion Focus
- 2 (Placebo Comparator): Group Psychotherapy- Self Esteem Focus
  Interventions: Behavioral: Group Psychotherapy- Self-Esteem Focus

INTERVENTIONS:
Behavioral: Group Psychotherapy-Negative Emotion Focus — 20 weekly sessions, 2 hours, group format
  Arms: 1
Behavioral: Group Psychotherapy- Self-Esteem Focus — 20 weekly sessions, 2 hours, group format
  Arms: 2

SUMMARY:
This study will compare two different approaches for the treatment for Binge Eating Disorder.

DETAILED DESCRIPTION:
Binge Eating Disorder (BED) is associated with impairments in physical, psychological, and social functioning. Research has revealed relationships between disordered eating and both low self-esteem and negative emotional states.

Participants in this study will complete assessment interviews regarding their eating disorder and associated problems. Similar assessments will be conducted at the end of the study. Participants will then be randomly assigned to one of two therapy groups. Participants in one group will focus on the role of self-esteem, self-awareness, and personal effectiveness in binge eating. Participants in the other group will focus on the role of negative emotions and binge eating. Both treatments will involve a 30 to 40 minute pre-treatment individual orientation session, followed by 20 weeks of weekly group therapy. Sessions will take place over 22 weeks, or approximately 6 months (18 weekly sessions followed by 2 biweekly sessions). Follow-up assessments will take place at 3 months, 6 months, and 12 months after study completion to assess maintenance of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Binge Eating Disorder
* Reside in the San Francisco Bay Area
* Willing to commit to the study requirements

Exclusion Criteria:

* Unstable medical problems
* History of bipolar illness or schizophrenia
* Receiving treatment for an eating disorder (or unwillingness to discontinue treatment upon study entry)
* Membership in weight-loss groups such as Weight Watchers or Jenny Craig (or unwillingness to discontinue membership upon study entry)
* Use of medications affecting weight or appetite. Antidepressants are acceptable, but doses of any psychiatric medication must have been stable for at least 3 months prior to study start
* Breast-feeding
* Require gastric-bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2003-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
frequency of binge eating | prior 4 weeks

SECONDARY OUTCOMES:
Emotional Eating Scale | prior 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Safer, MD, Principal Investigator — Stanford University Dept of Psychiatry
Locations (1):
- Stanford University Medical Center, Stanford, California, United States